CLINICAL TRIAL: NCT00633438
Title: A Double-Blind, Placebo-Controlled, Randomized Comparison Study of the Efficacy of Celebrex 400 mg Single Dose Pre and Celebrex 200 mg Post Ambulatory Arthroscopic Knee Surgery for Total Analgesic Use After Surgery
Brief Title: Effect of Celecoxib Versus Placebo Before and After Knee Surgery on Overall Use of Analgesics After Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A3191067
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Arthroscopy
Keywords: Knee Surgery Arthroscopic Surgery
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Placebo Comparator)
  Interventions: Other: Placebo
- A (Experimental)
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Other: Placebo — Matched oral capsule administered 1 hour prior to surgery and matched oral capsule administered post surgery as needed
  Arms: B
Drug: Celecoxib — 400 mg oral capsule as single dose administered 1 hour prior to surgery and 200 mg oral capsule as single dose administered post surgery as needed
  Arms: A

SUMMARY:
To compare total analgesic use at 24 hours after arthroscopic knee surgery in celecoxib-treated versus placebo-treated patients

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Diagnosed (or suspected to have) meniscus trauma of the knee requiring ambulatory arthroscopic knee surgery
* Willing to participate in study for 36 hours and come to follow-up visit 7 days post surgery

Exclusion Criteria:

Exclusion criteria:

* Osteoarthritis, inflammatory arthritis, or previous fracture of index joint
* Received acetaminophen or low dose narcotic (vicodin/tylox) within 8 hours of surgery
* Have received oral (4 weeks), intramuscular (2 months), intra-articular (3 months) or soft-tissue (2 months) injections of corticosteroids of the first dose of study medication or intra-artcular injections of hyaluronic acid in the index joint within 9 months of the first dose of study medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2004-01; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Total analgesic use (hydrocodone bitartrate 5 mg/acetaminophen 500 mg [HC/APAP]) after surgery | 24 hours

SECONDARY OUTCOMES:
Patient Assessment of Pain, according to visual analogue scale, after surgery at rest and flexion | 1, 2, 6, 8, 10, 12, 24, 36 hours
Time to analgesic use after surgery | 1, 2, 6, 8, 10, 12, 24, 36 hours
Number and percentage of patients taking HC/APAP after surgery | 1, 2, 6, 8, 10, 12, 24, 36 hours
Adverse events | Day 7
Physical exam | Day 7
Vital signs | Day 7
Laboratory evaluation | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (10):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Timonium, Maryland
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Orangeburg, South Carolina
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191067&StudyName=Effect%20of%20Celecoxib%20versus%20Placebo%20Before%20and%20After%20Knee%20Surgery%20on%20Overall%20Use%20of%20Analgesics%20After%20Surgery